CLINICAL TRIAL: NCT05647707
Title: The Efficacy of L-Carnitine in the Management of Acute Carbon Monoxide Poisoning
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, zahraa khalifa sobh, Associate Professor of Forensic Medicine and Clinical Toxicology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0304888
Record Dates: First submitted 2022-11-27; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Carbon Monoxide Poisoning
Keywords: Carbon Monoxide Poisoning; Cardiotoxicity; Troponin; L-Carnitine; Outcome
MeSH Terms: conditions — Carbon Monoxide Poisoning; Cardiotoxicity | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment randomized controlled clinical trial (phase II)
Who Masked: Outcomes Assessor
Masking Description: each patient will take a code number and data were analyzed anonymously
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Group (No Intervention): This group will comprise 36 patients who will receive conventional supportive treatment for the management of acute CO poisoning that include the following:
  * Airway: maintaining clear patent airways.
  * Breathing:
  * High-flow normobaric oxygen (NBO)
  * Hyperbaric oxygen (HBO) (if indicated).
  * Mechanical ventilation ( if required).
  * Circulation: intravenous fluids, and treatment of arrhythmias according to ECG abnormalities.
- L-Carnitine Group (Experimental): The 36 patients will receive conventional supportive care as in the conventional group in addition to IV L-carnitine.
  Interventions: Dietary Supplement: L-Carnitine

INTERVENTIONS:
Dietary Supplement: L-Carnitine — The 36 patients will receive conventional supportive care in addition to IV L-carnitine with a loading dose of 100 mg/kg IV over 30-60 min (maximum 6 g) and the maintenance dose of 50 mg/kg IV every 8 h.
  Arms: L-Carnitine Group

SUMMARY:
Carbon monoxide (CO) poisoning results in high morbidity and mortality worldwide. CO is described as a "silent killer" because CO is colorless, odorless, and tasteless but highly toxic. The diagnosis of acute CO poisoning depends on the history of exposure to a source of fire in a closed space along with the clinical and laboratory findings.

The pathophysiology of CO poisoning is not fully understood; however, it is proved that CO induces hypoxia by forming carboxyhemoglobin (COHb) and shifting the oxygen dissociation curve to the left. The molecular mechanisms of CO poisoning include oxidative injury through the generation of free radicals. In addition, oxygen therapy might enhance the reactive oxygen species (ROS) production and result in reperfusion injury. Free radicals could induce a serious impact on vital organs, including the heart, and brain.

L-Carnitine is an endogenous mitochondrial constituent that contributes to normal mitochondrial activities. L-Carnitine is an antioxidant with potent ROS scavenging ability. ROS-mediated pathology of CO suggests that antioxidants are potentially useful agents in the alleviation of CO toxicity. Thus, the current study will investigate the therapeutic efficacy of L-Carnitine in improving the prognosis of acute CO poisoning.

The current clinical trial will include patients with moderate and severe acute carbon monoxide poisoning according to Poisoning Severity Score.

DETAILED DESCRIPTION:
A randomized clinical trial (phase II) will be conducted at Alexandria Main University Hospital.

The total required sample size is 72. The sample size was calculated by G power 3.1.9.4 software program depending on the primary outcome. According to these assumptions: Effect size, defined as the difference between group 1 and group 2 in the mean troponin levels at 24 hr, was calculated according to Sun et al. (2011) and was 0.657, alpha error =0.05, power of 80%, allocation ratio 1:1. A 20% expected attrition was added to the sample size to account for loss to follow-up. So, the final sample size was 72; 36 patients per group.

All patients will be subject to the following:

1. History taking:

   * Personal data: age, and sex.
   * Exposure-related data: circumstances of exposure, and time till hospitalization.
   * Past medical history.
2. Clinical assessment:

   * Glasgow coma scale, vital signs, and general examination.
   * Laboratory investigations: arterial blood gases (ABG), Carboxy hemoglobin level (COHb), and cardiac enzymes (CPK, CK-MB, Troponin).
   * Electrocardiogram (ECG).

ELIGIBILITY:
Inclusion Criteria:

* The current clinical trials will include patients with moderate and severe acute carbon monoxide poisoning according to Poisoning Severity Score.

Exclusion Criteria:

* When the diagnosis of acute carbon monoxide poisoning is unconfirmed.
* Patients with advanced cardiac and neurological diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Troponin level | In follow-up 24 hours after admission
  Measure Troponin level in blood samples of patients

SECONDARY OUTCOMES:
Duration of hospital stay | Assessed up to 1 month.
  Time passed from the date of admission to the documented date of discharge or death, whichever came first
The frequency of ICU admission | Assessed up to 1 month.
  The number of patients admitted to ICU from the time of admission till the documented date of discharge or death, whichever came first. Patients who developed serious cardiovascular or neurological manifestations or need mechanical ventilation are indicated for ICU admission.
Development of delayed neurological manifestations | Assessed up to 3 months following discharge from the hospital
  The number of patients who developed impaired memory and or concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Zahraa K Sobh, MD, Principal Investigator — Associate Professor of Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Alexandria, Egypt; Maha A Ghanem, MD, Principal Investigator — Professor of Forensic Medicine and Clinical Toxicology. Head of department of Forensic Medicine and Clinical Toxicology. Chairperson of ethics committee Faculty of Medicine; Heidi A Elsobky, MS, Study Director — Assistant Lecturer of Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Alexandria, Egypt; Farah S Habib, Bachelor, Study Director — Demonstrator of Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Alexandria, Egypt; Fatma Elgazzar, MD, Principal Investigator — Professor of Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Tanta University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The confidentiality of the personal data of participants will be maintained. The current study will be published in an academic journal, then, the published data could be accessed and used for any purpose.

REFERENCES:
- [Background] Sun ZJ, Yang CB, Wang H, Li Y. [The impact of L-carnitine administration on the serum level of myocardium injury markers in patients with acute carbon monoxide poisoning]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2011 Dec;23(12):739-42. Chinese. PMID 22153012
- [Background] Zengin S, A B, Karta S, Can B, Orkmez M, Taskin A, Lok U, Gulen B, Yildirim C, Taysi S. An assessment of antioxidant status in patients with carbon monoxide poisoning. World J Emerg Med. 2014;5(2):91-5. doi: 10.5847/wjem.j.issn.1920-8642.2014.02.002. PMID 25215155
- [Background] Yildiz MN, Eroglu SE, Ozen C, Yildiz HA, Sektioglu BK, Alkan C. Analysis of the effects of COHb, lactate, and troponin levels on the clinical process and outcome in patients who were admitted to the emergency service due to carbon monoxide poisoning. North Clin Istanb. 2019 May 29;6(2):141-145. doi: 10.14744/nci.2018.88709. eCollection 2019. PMID 31297480
- [Background] Sherif NA, El-Banna AS, ElBourini MM, Khalil NO. Efficacy of L-carnitine and propranolol in the management of acute theophylline toxicity. Toxicol Res (Camb). 2020 Mar 11;9(1):45-54. doi: 10.1093/toxres/tfaa002. eCollection 2020 Feb. PMID 32440337
- [Background] Elgazzar FM, Elgohary MS, Basiouny SM, Lashin HI. Intravenous lipid emulsion as an adjuvant therapy of acute clozapine poisoning. Hum Exp Toxicol. 2021 Jul;40(7):1053-1063. doi: 10.1177/0960327120983873. Epub 2021 Jan 5. PMID 33401984